CLINICAL TRIAL: NCT02070497
Title: The Effectiveness of Nursing Case Management for Lung Cancer Patients in a Taiwan Medical Center
Brief Title: Effectiveness of Nursing Case Management for Lung Cancer Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 201005083R
Record Dates: First submitted 2012-11-19; First posted 2014-02-25 (Estimated); Last update posted 2014-02-25 (Estimated); Status verified 2014-02

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Case Management

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- case management_new (Experimental): The patients with new-diagnosed lung cancer and accepting case management
  Interventions: Other: case management
- case management_old (Experimental): the patients with non-new-diagnosed lung cancer and with accepting case management
  Interventions: Other: case management
- control group (No Intervention): The patients with new-diagnosed lung cancer in the period of one year ago and without accepting case management

INTERVENTIONS:
Other: case management — case management group will accept the case manager's service; the control group will just accept the routine care
  Other Names: nursing case management
  Arms: case management_new; case management_old

SUMMARY:
The study is to investigate the effectiveness of nursing case management for lung cancer patients in a Taiwan medical center.

DETAILED DESCRIPTION:
Purpose: The study is to investigate the effectiveness of nursing case management for lung cancer patients in a Taiwan medical center. The outcome variables include of percentages of patients accepted treatment in our medical center, average lengths of stay, unplanned re-admission rate, average admission times of emergency department per year, percentages of patients rejecting treatment, completing rate of treatment, withdrawing rate of treatment, improving rate of patients' treatment compliance, patients' satisfaction with healthcare, and staffs' satisfaction with case management.

Methods: The study will employ a quasi-experimental research design. The patients with new-diagnosed lung cancer and accepting case management will be assigned to the experimental group； The patients with new-diagnosed lung cancer in the period of one year ago and without accepting case management will be assigned to the control group；The third group is the patients with non-new-diagnosed lung cancer and with accepting case management. The staffs are the doctors within the lung cancer medical team.

The lung cancer case management database, patients' satisfaction questionnaire, and staffs' satisfaction questionnaire will be used to measure the effectiveness. Statistical software SPSS for Windows version 17.0 will be used to analyze the data.

Expected results: The research outcome will to confirm the impact of case management on the lung cancer patients and could be the reference data for future cancer case management model.

ELIGIBILITY:
Inclusion Criteria:

* patients with lung cancer

Exclusion Criteria:

* younger than 20 years old

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 415 (Actual)
Dates: Start 2010-07; Primary Completion 2011-08 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
chart review | One year
  We reviewed the chart and lung cancer case management database to collect the patients' healthy outcome. The outcome variables include of percentages of patients accepted treatment in our medical center, average lengths of stay, unplanned re-admission rate, average admission times of emergency department per year, percentages of patients rejecting treatment, completing rate of treatment, withdrawing rate of treatment, improving rate of patients' treatment compliance.

SECONDARY OUTCOMES:
patients' satisfaction questionnaire | 1 day
staffs' satisfaction questionnaire | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Ming-Ying Hong, RN, Master, Study Chair — Department of Nursing, National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital Research Ethics Committee, Taipei, Taipei, Taiwan